CLINICAL TRIAL: NCT05726539
Title: The Military Spouse Resiliency Group (MSRG) Peer Support Program: Equipping Families For Resiliency With Tools (EFFRT)
Brief Title: The Military Spouse Resiliency Group (MSRG) Peer Support Program: Equipping Families For Resiliency With Tools
Acronym: (EFFRT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00003159
Record Dates: First submitted 2023-01-02; First posted 2023-02-14 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Military Family
Keywords: military spouse; peer support; quality of life; social support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): participants receive group-based peer support
  Interventions: Behavioral: Group-based peer support
- Waitlist (No Intervention): participants wait to receive peer support until pre and post assessments are complete with their matched intervention group

INTERVENTIONS:
Behavioral: Group-based peer support — Receipt of semi-structured curriculum based group peer support that addresses common concerns of military spouses
  Arms: Intervention

SUMMARY:
This study will adapt and test an established peer support program for military spouses that offers them significant weekly group-based support on an array of topics that affect their lives. The curriculum will be able to be used in-person through group meetings or virtually by using a web-based meeting platform. The near-term impact of this study is that scientific knowledge will be developed about how well a curriculum-based, weekly, in-person support group for military spouses is effective in improving spouses' quality of life, mental health, social support and knowledge of health conditions impacting service members.

This study will assess whether offering military spouses support for coping with their mental health and social support needs to achieve a greater quality of life, a greater sense of social support and knowledge about and access to resources to address a range of issues they may be facing throughout their spouses' military careers. By educating them about the health conditions their service members may experience and how to support their recovery and access to treatment, service members will also benefit by having more familial support for seeking treatment. Educating family members about the injuries that SMs face will help to maintain stronger family relationships and reduce family relationship stress.

DETAILED DESCRIPTION:
This study will examine the impact of structured, evidence-based peer support group adapted to address the specific concerns of military spouses designed to increase social support, reduce depression and increase knowledge of SM health needs. Research Plan: This study will address Specific Aim 1:To adapt an existing veteran spouse peer support curriculum for active-duty spouses based on data collected from focus groups and interviews with military spouses, and Specific Aim 2: Conduct a randomized controlled trial (N = 150) to evaluate how military spouses' participation in a peer support group influences their mental health, quality of life and social support outcomes as well as improves their knowledge about psychological health problems faced by SMs and their confidence in supporting SM access to treatment. Hypothesis 1: Military spouses and significant others who participate in the Military Spouse Resiliency Group (M-SRG) program will show improved quality of life, sense of social support, self-care practices and depression symptoms.Hypothesis 2: After completing M-SRG participants will possess greater knowledge of common SM psychological health problems and greater confidence in how to support SMs' access to care.Impact: The near-term impact of this study and its products are that scientific knowledge will be developed about how well a curriculum-based, weekly, in-person support group for military spouses is effective in improving spouses' quality of life, mental health, social support and knowledge of health conditions impacting service members. The long-term impact of this study will be to offer ongoing, necessary health and social support to spouses through peer support groups. Equipping spouses with skills to address the mental health and healthcare needs of SMs will provide spouses necessary supports for their unique experiences as part of military life.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be married to or in a committed relationship with a service member stationed at Fort Hood;
* Participants must have a reasonable expectation of remaining at Fort Hood for at least 4 months.
* Participants must be willing to attend up to 10 sessions of a military spouse peer support group in person at Fort Hood.

Exclusion Criteria:

* Spouses who are separated or divorced from a service member are not eligible to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-05 (Estimated); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire (Short Form) (Q-LES-Q-SF) | Change in Quality of Life Enjoyment and Satisfaction Questionnaire (Short Form) (Q-LES-Q-SF) from baseline, 2-weeks, 3 months
  The Quality of Life Enjoyment and Satisfaction Questionnaire measures satisfaction and enjoyment in different areas of daily functioning.
Patient Health Questionnaire-9 | Change in Patient Health Questionnaire-9 from baseline, 2-weeks, and 3-months
  The Patient Health Questionnaire-9 measures symptoms of depression.
Military Spouse Self-Care Inventory (MSSCI) | Change in Military Spouse Self-Care Inventory from baseline, 2-weeks, and 3-months
  The Military Spouse Self-Care Inventory assesses five domains of self-care that military spouses regularly practice.
Interpersonal Support Evaluation List-12 (ISEL-12) | Change in Interpersonal Support Evaluation List-12 from baseline, 2-weeks, and 3-months
  The Interpersonal Support Evaluation List-12 is used to measure perceived social support. It has been widely used (Donoho et al., 2017) as a short-form measure of the traditional ISEL, which measures perceived social support (Cohen et al., 1985).
Psychological Health Knowledge Assessment | Change in Psychological Health Knowledge Assessment from baseline, 2-weeks, and 3-months
  Investigator-developed assessment of common psychological health concerns and available treatments commonly affecting service members
General Anxiety Disorder-7 (GAD-7) | Change in General Anxiety Disorder-7 from baseline, 2-weeks, and 3-months
  General Anxiety Disorder-7 is a valid and reliable instrument to measure generalized anxiety (Spitzer et al., 2006). Minimum is 0 and maximum is 21 and higher scores indicate more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Borah, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow JH, Turner AP, Wright CC. A randomized controlled study of the Arthritis Self-Management Programme in the UK. Health Educ Res. 2000 Dec;15(6):665-80. doi: 10.1093/her/15.6.665. PMID 11142075
- [Background] Campbell SB, Renshaw KD. PTSD symptoms, disclosure, and relationship distress: explorations of mediation and associations over time. J Anxiety Disord. 2013 Jun;27(5):494-502. doi: 10.1016/j.janxdis.2013.06.007. Epub 2013 Jul 9. PMID 23917126
- [Background] Donoho CJ, LeardMann C, O'Malley CA, Walter KH, Riviere LA, Curry JF, Adler AB. Depression among military spouses: Demographic, military, and service member psychological health risk factors. Depress Anxiety. 2018 Dec;35(12):1137-1144. doi: 10.1002/da.22820. Epub 2018 Aug 13. PMID 30103266
- [Background] Eaton KM, Hoge CW, Messer SC, Whitt AA, Cabrera OA, McGurk D, Cox A, Castro CA. Prevalence of mental health problems, treatment need, and barriers to care among primary care-seeking spouses of military service members involved in Iraq and Afghanistan deployments. Mil Med. 2008 Nov;173(11):1051-6. doi: 10.7205/milmed.173.11.1051. PMID 19055177
- [Background] Griffiths C, Motlib J, Azad A, Ramsay J, Eldridge S, Feder G, Khanam R, Munni R, Garrett M, Turner A, Barlow J. Randomised controlled trial of a lay-led self-management programme for Bangladeshi patients with chronic disease. Br J Gen Pract. 2005 Nov;55(520):831-7. PMID 16281998
- [Background] Humphreys K, Wing S, McCarty D, Chappel J, Gallant L, Haberle B, Horvath AT, Kaskutas LA, Kirk T, Kivlahan D, Laudet A, McCrady BS, McLellan AT, Morgenstern J, Townsend M, Weiss R. Self-help organizations for alcohol and drug problems: toward evidence-based practice and policy. J Subst Abuse Treat. 2004 Apr;26(3):151-8; discussion 159-65. doi: 10.1016/S0740-5472(03)00212-5. PMID 15063905
- [Background] Kees M, Rosenblum K. Evaluation of a psychological health and resilience intervention for military spouses: A pilot study. Psychol Serv. 2015 Aug;12(3):222-30. doi: 10.1037/ser0000035. PMID 26213791
- [Background] Kennedy A, Reeves D, Bower P, Lee V, Middleton E, Richardson G, Gardner C, Gately C, Rogers A. The effectiveness and cost effectiveness of a national lay-led self care support programme for patients with long-term conditions: a pragmatic randomised controlled trial. J Epidemiol Community Health. 2007 Mar;61(3):254-61. doi: 10.1136/jech.2006.053538. PMID 17325405
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Lester P, Peterson K, Reeves J, Knauss L, Glover D, Mogil C, Duan N, Saltzman W, Pynoos R, Wilt K, Beardslee W. The long war and parental combat deployment: effects on military children and at-home spouses. J Am Acad Child Adolesc Psychiatry. 2010 Apr;49(4):310-20. PMID 20410724
- [Background] Long JA, Jahnle EC, Richardson DM, Loewenstein G, Volpp KG. Peer mentoring and financial incentives to improve glucose control in African American veterans: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):416-24. doi: 10.7326/0003-4819-156-6-201203200-00004. PMID 22431674
- [Background] Mailey EL, Mershon C, Joyce J, Irwin BC. "Everything else comes first": a mixed-methods analysis of barriers to health behaviors among military spouses. BMC Public Health. 2018 Aug 15;18(1):1013. doi: 10.1186/s12889-018-5938-z. PMID 30111307
- [Background] Pfeiffer PN, Heisler M, Piette JD, Rogers MA, Valenstein M. Efficacy of peer support interventions for depression: a meta-analysis. Gen Hosp Psychiatry. 2011 Jan-Feb;33(1):29-36. doi: 10.1016/j.genhosppsych.2010.10.002. Epub 2010 Nov 13. PMID 21353125
- [Background] Pflieger JC, LeardMann CA, McMaster HS, Donoho CJ, Riviere LA; Millennium Cohort Family Study Team. The Impact of Military and Nonmilitary Experiences on Marriage: Examining the Military Spouse's Perspective. J Trauma Stress. 2018 Oct;31(5):719-729. doi: 10.1002/jts.22321. Epub 2018 Oct 19. PMID 30338551
- [Background] Schulz U, Pischke CR, Weidner G, Daubenmier J, Elliot-Eller M, Scherwitz L, Bullinger M, Ornish D. Social support group attendance is related to blood pressure, health behaviours, and quality of life in the Multicenter Lifestyle Demonstration Project. Psychol Health Med. 2008 Aug;13(4):423-37. doi: 10.1080/13548500701660442. PMID 18825581
- [Background] Solomon P. Peer support/peer provided services underlying processes, benefits, and critical ingredients. Psychiatr Rehabil J. 2004 Spring;27(4):392-401. doi: 10.2975/27.2004.392.401. PMID 15222150
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Steenkamp MM, Corry NH, Qian M, Li M, McMaster HS, Fairbank JA, Stander VA, Hollahan L, Marmar CR. Prevalence of psychiatric morbidity in United States military spouses: The Millennium Cohort Family Study. Depress Anxiety. 2018 Sep;35(9):815-829. doi: 10.1002/da.22768. Epub 2018 May 10. PMID 29745445
- [Background] Stevanovic D. Quality of Life Enjoyment and Satisfaction Questionnaire-short form for quality of life assessments in clinical practice: a psychometric study. J Psychiatr Ment Health Nurs. 2011 Oct;18(8):744-50. doi: 10.1111/j.1365-2850.2011.01735.x. Epub 2011 May 5. PMID 21896118